CLINICAL TRIAL: NCT03613987
Title: Randomized Control Trial: Synchronized Non-Invasive Positive Pressure Ventilation (sNIPPV) With Neurally-Assisted Ventilatory Assist (NAVA) Versus NIPPV in Extremely Low Birth Weight Infants
Brief Title: Randomized Control Trial: Synchronized Non-invasive Positive Pressure Ventilation Versus Non Synchronized Non Invasive Positive Pressure Ventilation in Extremely Low Birth Weight Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: L12,175
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: BPD - Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NIPPV (No Intervention): non synchronized non invasive positive pressure ventilation
- NAVA-NIPPV (Experimental): synchronized non invasive positive pressure ventilation with NAVA
  Interventions: Device: NAVA technology to synchronize NIPPV

INTERVENTIONS:
Device: NAVA technology to synchronize NIPPV — Neurally adjust ventilator assist is used to synchronize the NIPPV
  Arms: NAVA-NIPPV

SUMMARY:
Infants delivered weighing less than 1 kg at birth (ELBW) are at high risk for the development of bronchopulmonary dysplasia (BPD) and Ventilator-Induced Lung Injury (VILI), in part because of the need for mechanical ventilation utilizing an endotracheal tube (MVET). In spite of strategies to minimize the need for MVET, the incidence of BPD in ELBW infants continues to be 20-80%. The hypothesis is that synchronized NIPPV will decrease the need for MVET and reduce BPD in ELBW infants as compared to NIPPV.

DETAILED DESCRIPTION:
Hypothesis:

The hypothesis is that sNIPPV will decrease the need for MVET and reduce BPD in ELBW infants as compared to NIPPV.

Specific Aims:

The specific aims are to determine whether:

1. sNIPPV results in a decreased need for MVET at 7days of life and 28 days of life in ELBW infants compared to NIPPV.
2. sNIPPV reduces BPD in ELBW infants compared to NIPPV. Research design and methods: ELBW infants will be enrolled in this study at the RNICU at MFCH of WMC following informed written parental consent.

Randomization:

ELBW infants will be randomized to either sNIPPV group or NIPPV group using a computer-generated scheme.

Extubation criteria:

1. Infant is receiving caffeine.
2. Infants can be extubated at any point, but must be extubated following a 12-hour period of clinical stability when the ventilator settings have met all the following criteria:

   * mean airway pressure (MAP) < 8cmH20,
   * FiO2 < 0.4,
   * pH > 7.2, and
   * pCO2 < 70.

Intubation criteria:

Infants must be intubated if any of the following criteria occur:

1. One apneic event requiring positive pressure ventilation (PPV).
2. More than 6 apneic events requiring stimulation within a 6-hour period.
3. A deterioration in respiratory status as noted by any of the following criteria:

   * pH < 7.2,
   * pCO2 > 70,
   * FiO2 > 0.6,
4. Or, if in the opinion of the attending neonatologist, the baby is failing either non-invasive strategy.

Data Collection:

Demographic and outcome data will be collected from source data, and then the patient will be given a unique identifier, without reference to MRN or birthdate.

Tracheal aspirates will be collected per routine nursing care to look for inflammatory cytokine markers (IL8, IL6 and TNF alpha). This may help to determine if certain infants remained intubated due to a pro-inflammatory mechanism (if their TA cytokines were elevated early compared to those who may have been more successfully extubated because of low levels of cytokines).

During hospital stay, DNA and RNA samples will be extracted from buccal swabs, as certain babies are more susceptible to BPD based on their genetic foundations.

Charts will be reviewed to determine the duration of oxygen therapy as well as the duration of MVET.

MVET will be assessed at 7 days of life and 28 days of life as primary outcome. BPD, as defined as oxygen requirement at 36 weeks PMA, is a secondary outcome. Initial statistical analysis will be performed using chi square for categorical data; and t-test or Mann Whitney for continuous data that is normally or non-normally distributed (respectively), with statistical significance when P < 0.05.

Power analysis:

Based on the investigators' NICU data that NIPPV has MVET rate at 7 days of life of 84% for ELBWs, it was hypothesized that sNIPPV will decrease the need for MVET at 7 days of life by 40%. For a power of 80%, and an alpha value of 0.05, the sample size is 27 infants in each group. Anticipating a 10% dropout rate, this gives 30 as the sample size for each group.

Anticipated timeline:

With 80-100 ELBW infants admitted each year, enrollment is anticipated to be completed in 1 year.

The clinical implications of this study will determine if synchronized NIPPV in ELBW infants will reduce the need for mechanical ventilation and ultimately BPD.

There are no procedures, situations, or materials that will be hazardous to personnel. There are no courses planned which support the research training experience. This research will not include the use of experimental drugs or treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Babies born less than 1kg.
2. Babies born at 24-30 weeks gestation.
3. Babies who qualify for surfactant administration within 90mins of birth:

   * FiO2 > 0.4,
   * nCPAP > 6, with
   * Increased work of breathing as noted by grunting; and/or inter-, sub-, or supra-sternal retractions.

Exclusion Criteria:

1. Babies with Grade 3-4 IVH (may not be known prior to randomization).
2. Babies with congenital anomalies including neuromuscular disorder.
3. Babies who do not require intubation until 7 days of life.

Ages: 24 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

PRIMARY OUTCOMES:
The need for Mechanical Ventilation via ET tube ( MVET) at 7 days of life | 7 days of life
  Mechanical ventilation via Endotracheal tube
The need for Mechanical Ventilation via ET tube ( MVET) at 28 days of life | 28 days of life
  Mechanical Ventilation via Endotracheal tube

SECONDARY OUTCOMES:
Incidence of BPD or need for supplemental O2 at 36 weeks corrected age | 36 weeks corrected gestational age
  Bronchopulmonary Dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Lance Parton, MD, Principal Investigator — Westchester Medical Center
Locations (1):
- Westchester Medical Center, Valhalla, New York, United States

REFERENCES:
- [Derived] Louie K, Amatya S, Alpan G, Parton LA. Non-Invasive Ventilation with Neurally Adjusted Ventilatory Assist (NAVA) Improves Extubation Outcomes in Extremely Low-Birth-Weight Infants. Children (Basel). 2024 Sep 28;11(10):1184. doi: 10.3390/children11101184. PMID 39457149